CLINICAL TRIAL: NCT02831127
Title: Mobile Phone Reminder Messages Improves the Adherence of Stent Removal or Exchange in Patients With Benign Pancreaticobiliary Diseases
Brief Title: Mobile Messages Affects Adherence of Stent Removal or Exchange in Patients With Benign Pancreaticobiliary Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20160707-1
Record Dates: First submitted 2016-07-10; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: short message service; adherence; stent exchange; ERCP

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- short message service group (Experimental): Patients in this arm received conventional instructions plus short message reminder.
  Interventions: Other: short message service group
- conventional group (Active Comparator): Patients in this arm just received conventional instructions.
  Interventions: Other: conventional group

INTERVENTIONS:
Other: short message service group — Each month after stent implantation, the investigator sent a text message by SMS to inform patients the necessity of regular stent removal/exchange and the disadvantage of delayed management, and to remind them the appropriate date to come back to the hospital for stent management. Patients were requested to respond by SMS and were encouraged to contact the investigator if they had any questions about stent management. Besides, patients received conventional reminder:After stent implantation, all patients received oral and written instructions about further management. If single or multiple plastic stents were inserted, patients were informed to come back to the hospital at 3 months for stent removal/exchange; if FCSEMS was inserted, they were informed to come back to the hospital at 6 months after ERCP.
  Arms: short message service group
Other: conventional group — After stent implantation, all patients received oral and written instructions about further management. If single or multiple plastic stents were inserted, patients were informed to come back to the hospital at 3 months for stent removal/exchange; if FCSEMS was inserted, they were informed to come back to the hospital at 6 months after ERCP.
  Arms: conventional group

SUMMARY:
Plastic and covered metal stents need to be removed or exchanged within appropriate time in case of undesirable complications. However, it is not uncommon that patients does not follow the recommendation for further stent management after ERCP. we hopothesized that short message service (SMS) intervention monthly could improve the adherence in patients with benign pancreaticobiliary after ERCP.

ELIGIBILITY:
Inclusion Criteria:

* be able to communicate via SMS by mobile phones of themselves or relatives living together

Exclusion Criteria:

* primary or secondary sclerosing cholangitis (PSC)
* malignant or suspected malignant stricture of biliary or pancreatic duct
* implantation of pancreatic duct (PD) stent for prevention of post-ERCP pancreatitis
* expected survival time less than 6 months
* plan of surgery within 6 months
* pregnant or lactating women
* patients who could not give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Adherence rate of biliary stent removal/exchange | up to 1 year
  Percentage of patients adherence to stent removal/exchange within appropriate time

SECONDARY OUTCOMES:
Stent-associated adverse event | 1 year
  Percentage of patients with stent-related adverse events, including cholangitis, stent migration and abdominal pain

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, MD, Principal Investigator — Xijing Hospital of Disgestive Diseases.The Fourth Military University
Locations (1):
- Endoscopic center, Xijing Hospital of Digestive Diseases, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gu Y, Wang L, Zhao L, Liu Z, Luo H, Tao Q, Zhang R, He S, Wang X, Huang R, Zhang L, Pan Y, Guo X. Effect of mobile phone reminder messages on adherence of stent removal or exchange in patients with benign pancreaticobiliary diseases: a prospectively randomized, controlled study. BMC Gastroenterol. 2016 Aug 26;16(1):105. doi: 10.1186/s12876-016-0522-4. PMID 27565717